CLINICAL TRIAL: NCT05360875
Title: The Effect of Endometrial Scratching on Patients With Endometriosis Undergoing IVF Treatment
Brief Title: The Effect of Endometrial Scratching on Patients With Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qi Yu, professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2065
Record Dates: First submitted 2022-05-01; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis; IVF
Keywords: Endometriosis; Endometrial scratching; Endometrial receptivity; IVF; Pregnancy rates
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrial scratching group (Experimental)
  Interventions: Procedure: Endometrial scratching
- Non-scratching group (No Intervention)

INTERVENTIONS:
Procedure: Endometrial scratching — An intrauterine procedure that causes mild endometrial injury
  Arms: Endometrial scratching group

SUMMARY:
We aimed to investigate whether endometrial scratching could improve IVF outcomes by enhancing endometrial receptivity in patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

1.Endometriosis that surgery or pathology confirmed; 2. normal ovarian reserve; 3. at least one implantation failure history

Exclusion Criteria:

1. hydrosalpinx; 2.ademomyosis; 3.endocrine or self-immune disease; 4.serious medical condition; 5.Contraindications of intrauterine operation

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 6-7 weeks of gestation
  pregnancy sacs confirmed by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol